CLINICAL TRIAL: NCT00774098
Title: Improving Glycogen Liver Content Will Improve Post-operative Liver Function in Patients Undergoing Major Liver Resections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Dr Peter Metrakos, MUHC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SDR-06-012
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: Liver Function
Keywords: all adult patients (>18 years) planned to undergo a major liver resection
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Intravenous normal saline (NS 0.9) started just before induction, and titrated to hemodynamic parameters and urine output
  Interventions: Drug: Intravenous normal saline (NS 0.9)
- GICP (Experimental)
  Interventions: Drug: dextrose 10% (D10W ®) infusion; Drug: hyperinsulinemic normoglycemic clamp; Dietary Supplement: high calorie diet 35 kcal/kg

INTERVENTIONS:
Drug: dextrose 10% (D10W ®) infusion — Started at 8pm the day before surgery until the procedure begins
  Arms: GICP
Drug: hyperinsulinemic normoglycemic clamp — Started as the procedure begins, decreased at the end of the procedure and continued until 16 hours postoperatively
  Arms: GICP
Dietary Supplement: high calorie diet 35 kcal/kg — High Calorie meals start the day before the surgery and are given 5 hours apart. The last meal is given at 7 pm the day before surgery
  Arms: GICP
Drug: Intravenous normal saline (NS 0.9) — Intravenous normal saline (NS 0.9) started just before induction, and titrated to hemodynamic parameters and urine output
  Arms: Control Group

SUMMARY:
We would like to study the effect of preserving liver glycogen storage by using intravenous dextrose infusion on postoperative liver function and complications after major liver resections.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* planned to undergo a major liver resection at McGill University Health Center (MUHC)

Exclusion Criteria:

* patients known with chronic viral liver disease
* uncontrolled or type one diabetes mellitus (DM)
* patients on oral beta-blocker agents
* patients with unresectable disease determined intra-operatively
* patients unable to give consent for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Postoperative liver function test | Postoperative

SECONDARY OUTCOMES:
Liver and muscle glycogen, TG, and protein content at beginning and end of the procedure. | Begining + end of the procedure
Incidence of complications | Postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Hassanain M, Metrakos P, Fisette A, Doi SA, Schricker T, Lattermann R, Carvalho G, Wykes L, Molla H, Cianflone K. Randomized clinical trial of the impact of insulin therapy on liver function in patients undergoing major liver resection. Br J Surg. 2013 Apr;100(5):610-8. doi: 10.1002/bjs.9034. Epub 2013 Jan 21. PMID 23339047
- [Derived] Fisette A, Hassanain M, Metrakos P, Doi SA, Salman A, Schricker T, Lattermann R, Wykes L, Nitschmann E, Smith J, Cianflone K. High-dose insulin therapy reduces postoperative liver dysfunction and complications in liver resection patients through reduced apoptosis and altered inflammation. J Clin Endocrinol Metab. 2012 Jan;97(1):217-26. doi: 10.1210/jc.2011-1598. Epub 2011 Oct 26. PMID 22031518
- [Derived] Sato H, Lattermann R, Carvalho G, Sato T, Metrakos P, Hassanain M, Matsukawa T, Schricker T. Perioperative glucose and insulin administration while maintaining normoglycemia (GIN therapy) in patients undergoing major liver resection. Anesth Analg. 2010 Jun 1;110(6):1711-8. doi: 10.1213/ANE.0b013e3181d90087. Epub 2010 Apr 7. PMID 20375299